CLINICAL TRIAL: NCT03181971
Title: The Impact of the School Water Access on Child Food and Beverage Intake and Obesity
Brief Title: School Water Access, Food and Beverage Intake, and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); University of California (Other)
Responsible Party: Principal Investigator, Anisha I Patel, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL129288-01A1 (NIH)
Record Dates: First submitted 2017-06-03; First posted 2017-06-09 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: water; sugar-sweetened beverages; schools
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water Access and Promotion - Students (Experimental): Intervention group will receive installation of water stations in high traffic areas, schoolwide promotion, and 4th graders will receive a curricula focused on increasing intake of water.
  Interventions: Behavioral: Water First
- Control - Students (No Intervention): Participants do not receive an intervention
- School Personnel (No Intervention): School administrators and food service managers provide information on school policies and procedures.

INTERVENTIONS:
Behavioral: Water First — The Water First intervention consists of increased access to safe and appealing drinking water in schools, school-wide promotion to increase students' intake of water, and education directed to 4th grade students and their families to increase intake of water.
  Arms: Water Access and Promotion - Students

SUMMARY:
It is widely argued that the promotion of water consumption, as an alternative to sugar-sweetened beverages, can assist in childhood obesity prevention efforts. Yet no studies have tested this argument in real world schools where flavored milk or juices are available. This trial will fill gaps by examining how promoting fresh water intake-both in schools that do and do not provide access to caloric beverages -impacts children's consumption of food and beverages both during and outside of school, and obesity.

DETAILED DESCRIPTION:
Maintaining a healthy weight is important for young children because childhood obesity is predictive of adult obesity and related chronic illness. Intake of sugar-sweetened beverages (SSBs: sodas, flavored milks, fruit-flavored drinks, and other drinks with added sugar) is a major contributor to obesity. This is particularly true for low income children who are more likely to drink SSBs and to be obese. Children spend substantial time in schools where they consume up to 50% of daily calories, including those from SSBs. Consequently, many obesity prevention efforts have targeted reductions in SSB intake in schools. Recently, scientific authorities have also recommended that schools improve the availability of potable and free drinking water - a healthy alternative to SSBs - as a low-cost and feasible obesity prevention strategy. Emerging policies also mandate water access in schools; but implementation is poor. Although the 2010 Healthy, Hunger-Free Kids Act requires schools participating in federal meal programs to provide free potable water where meals are served, 25% of US schools still fail to do so. And even in schools that offer free water, drinking fountains may be avoided due to concerns about cleanliness or sub-standard water quality. While promotion of drinking water intake in schools is a plausible obesity prevention strategy, no large studies have systematically examined how this tactic can change children's overall dietary patterns and obesity rates in schools that offer SSBs and juices. This study's central hypothesis is that in elementary schools, increased access to fresh water and rigorous promotion of its consumption will reduce student intake of caloric beverages, thereby leading to lower rates of obesity. This hypothesis will be tested through a cluster-randomized trial in 26 low-income elementary schools in the San Francisco Bay Area, in which 13 schools will receive a water promotion intervention and 13 schools will serve as controls. The intervention, based on Social Cognitive Theory and the PRECEDE-PROCEED Model and cultivated in the investigators' prior developmental studies, promotes water consumption by: 1) installing lead-free water stations in cafeterias, physical activity spaces and high-traffic common areas, 2) providing cups and reusable water bottles for students, and 3) conducting a 6-month health education campaign that includes a kick-off play, class lessons, family homework activities, signage, and rewards. From baseline to 7 and 15 months after the start of the intervention, researchers measure differences in: 1) water intake (observations and measurements of water taken from water sources) 2) water and SSB intake via beverage frequency questionnaires and 3) overweight/obesity prevalence between students in intervention and control schools. Total caloric intake from foods and beverages (24-hour food and beverage diaries) are measured at baseline and 7 months only due to budget cuts and their resource intensiveness. If the proposed school water intervention is effective, school officials will have a feasible and low-cost obesity prevention tool. US schools will soon be federally mandated to reevaluate their wellness policies in order to implement new food and beverage regulations. This study presents a timely opportunity to provide leaders with an evidence-based strategy for improving student nutrition and health.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade students, students in 4th grade combination classes who speak English or Spanish and who don't have health conditions that preclude intake of water
* School administrators and food service directors at study schools

Exclusion Criteria:

* Students not in the 4th grade or 4th grade combination classes
* Students who do not speak English or Spanish

Ages: 9 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1861 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Patel, MD, MSPH, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezennia J, Schmidt LA, Ritchie LD, Blacker L, McCulloch CE, Patel AI. Water Security Experiences and Water Intake Among Elementary Students at Low-Income Schools: A Cross-Sectional Study. Acad Pediatr. 2023 Jan-Feb;23(1):68-75. doi: 10.1016/j.acap.2022.04.008. Epub 2022 May 7. PMID 35537674
- [Background] Moreno GD, Schmidt LA, Ritchie LD, McCulloch CE, Cabana MD, Brindis CD, Green LW, Altman EA, Patel AI. A cluster-randomized controlled trial of an elementary school drinking water access and promotion intervention: Rationale, study design, and protocol. Contemp Clin Trials. 2021 Feb;101:106255. doi: 10.1016/j.cct.2020.106255. Epub 2020 Dec 25. PMID 33370616
- [Result] Patel AI, Schmidt LA, McCulloch CE, Blacker LS, Cabana MD, Brindis CD, Ritchie LD. Effectiveness of a School Drinking Water Promotion and Access Program for Overweight Prevention. Pediatrics. 2023 Sep 1;152(3):e2022060021. doi: 10.1542/peds.2022-060021. PMID 37545466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cluster-randomized trial: participants were enrolled from schools that were randomized to receive the intervention, or no intervention.
Pre-assignment Details: 1861 students and adults signed consent; 564 students and adults could not be in the study due to pandemic school closures.
Units Other Than Participants: Schools
Groups:
- Water Access and Promotion - Students: Schools receive installation of water stations in high traffic areas, schoolwide promotion, and 4th graders receive a curricula focused on increasing intake of water (intervention group). School personnel complete surveys on school policies and procedures.
- Control - Students: Schools do not receive the intervention. School personnel complete surveys on school policies and procedures.
- Food Service Directors: District-level Food Service Directors complete surveys on school policies and procedures.
Period: Overall Study
Arm/Group | Water Access and Promotion - Students | Control - Students | Food Service Directors
Started | 690; 9 Schools | 594; 9 Schools | 13; 0 Schools
Students Who Started the Study | 680; 9 Schools | 582; 9 Schools | 0; 0 Schools
Adults Who Started Study | 10; 9 Schools | 12; 9 Schools | 13; 0 Schools
Students That Received Allocated Intervention / Participated in Allocated Control | 677; 9 Schools | 572; 9 Schools | 0; 0 Schools
Students Who Completed the Study | 548; 9 Schools | 510; 9 Schools | 0; 0 Schools
Adults Who Completed the Study | 10; 9 Schools | 12; 9 Schools | 13; 0 Schools
Completed | 558; 9 Schools | 522; 9 Schools | 13; 0 Schools
Not Completed | 132; 0 Schools | 72; 0 Schools | 0; 0 Schools

BASELINE CHARACTERISTICS:
Population: Student who received allocated intervention or participated in allocated control, and adult participants.
Groups:
- Water Access and Promotion - Students: Schools receive installation of water stations in high traffic areas, schoolwide promotion, and 4th graders receive a curricula focused on increasing intake of water (intervention group).
- Water Access and Promotion - School Personnel: Schools receive installation of water stations in high traffic areas, schoolwide promotion (intervention group). School personnel complete surveys on school policies and procedures.
- Control - Students: Schools do not receive an intervention.
- Control - School Personnel: Schools do not receive an intervention. School personnel complete surveys on school policies and procedures.
- Total: Total of all reporting groups
Arm/Group | Water Access and Promotion - Students | Water Access and Promotion - School Personnel | Control - Students | Control - School Personnel | Food Service Directors | Total
Number analyzed (Participants) | 677 | 10 | 572 | 12 | 13 | 1284
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data were not gathered from the adult participants.
  years
    number analyzed (Participants) | 677 | 0 | 572 | 0 | 0 | 1249
    (all) | 9.6 (0.4) |  | 9.6 (0.4) |  |  | 9.6 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 318 | 5 | 274 | 6 | 13 | 616
  Male | 359 | 5 | 298 | 6 | 0 | 668
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/ethnicity data were not gathered from the adult participants.
  Participants
    Race and ethnicity, No (%): number analyzed (Participants) | 677 | 0 | 572 | 0 | 0 | 1249
    Race and ethnicity, No (%): Mexican American, Latino, Hispanic | 455 |  | 337 |  |  | 792
    Race and ethnicity, No (%): Non-Hispanic Asian | 80 |  | 94 |  |  | 174
    Race and ethnicity, No (%): Non-Hispanic Black | 26 |  | 25 |  |  | 51
    Race and ethnicity, No (%): Non-Hispanic White | 43 |  | 45 |  |  | 88
    Race and ethnicity, No (%): Other (including American Indian or Alaska Native) | 73 |  | 71 |  |  | 144
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 677 | 10 | 572 | 12 | 13 | 1284

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Age- and Sex-adjusted BMI% Greater Than or Equal to 85%
Description: Trained research staff will measure students' heights and weights as outlined in the National Health and Nutrition Examination Survey Anthropometry Procedures Manual.
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: Outcome measure data were collected from students only. Participants with data at each respective time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Water Access and Promotion - Students: Intervention group receives installation of water stations in high traffic areas, schoolwide promotion, and 4th graders receive a curricula focused on increasing intake of water.
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 677 | 572
Participants
  Baseline | 335 | 273
  Month 7: number analyzed (Participants) | 639 | 556
  Month 7 | 315 | 263
  Month 15: number analyzed (Participants) | 548 | 510
  Month 15 | 274 | 262
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 7 months; Test type: Superiority; p = 0.68, Mixed Models Analysis; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.2 to 2.9]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 15 months; Test type: Superiority; p = 0.017, Mixed Models Analysis; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.03 to 0.7]

2. Secondary Outcome: Number of Participants With Age- and Sex-adjusted BMI% Greater Than or Equal to 95%. Yes or No.
Description: as for outcome 1
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 677 | 572
Participants
  Baseline | 222 | 165
  Month 7: number analyzed (Participants) | 639 | 556
  Month 7 | 202 | 159
  Month 15: number analyzed (Participants) | 548 | 510
  Month 15 | 179 | 144
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 7 months; Test type: Superiority; p = .24, Mixed Models Analysis; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.07 to 2.0]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 15 months; Test type: Superiority; p = .98, Mixed Models Analysis; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.1 to 7.0]

3. Secondary Outcome: BMI Percentile,Mean(SD)
Description: as for outcome 1
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BMI-for-age/sex percentile
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 677 | 572
BMI-for-age/sex percentile
  Baseline | 73.2 (28.1) | 71.9 (28.7)
  Month 7: number analyzed (Participants) | 639 | 556
  Month 7 | 73.7 (27.1) | 71.8 (28.4)
  Month 15: number analyzed (Participants) | 548 | 510
  Month 15 | 73.5 (28.0) | 72.9 (28.5)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 7 months; Test type: Superiority; p = 0.57, Mixed Models Analysis; Adjusted mean difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 15 months; Test type: Superiority; p = .40, Mixed Models Analysis; Adjusted mean difference = -0.5, 95% CI 2-sided [-1.5 to 0.6]

4. Secondary Outcome: BMI, Mean (SD)
Description: as for outcome 1
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 677 | 572
kg/m^2
  Baseline | 20.4 (4.6) | 20.1 (4.6)
  Month 7: number analyzed (Participants) | 639 | 556
  Month 7 | 20.9 (4.7) | 20.5 (4.7)
  Month 15: number analyzed (Participants) | 548 | 510
  Month 15 | 21.4 (5.1) | 21.2 (4.9)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 7 months; Test type: Superiority; p = .46, Mixed Models Analysis; Adjusted mean difference = 0.04, 95% CI 2-sided [-0.06 to 0.1]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 15 months; Test type: Superiority; p = .80, Mixed Models Analysis; Adjusted mean difference = -0.02, 95% CI 2-sided [-0.2 to 0.1]

5. Secondary Outcome: BMI Z-score, Mean (SD)
Description: Trained research staff will measure students' heights and weights as outlined in the National Health and Nutrition Examination Survey Anthropometry Procedures Manual. BMI z-scores (or standard deviation scores) are used in anthropometry to quantify a measurement's distance from the mean. The measurement is obtained using the sex, age, weight and height of the participants. The z-score is based on United States Centers for Disease Control and Prevention growth references for children. A z-score of 0 reflects the 50th percentile based on the reference growth charts. For example, a z-score of 1.5 indicates a child is 1.5 standard deviations above the average value, whereas a z-score of -1.5 means a child is 1.5 standard deviations below the average value.
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 677 | 572
z-score
  Baseline | 0.9 (1.1) | 0.8 (1.1)
  Month 7: number analyzed (Participants) | 639 | 556
  Month 7 | 0.9 (1.1) | 0.8 (1.1)
  Month 15: number analyzed (Participants) | 548 | 510
  Month 15 | 0.9 (1.1) | 0.9 (1.1)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 7 months; Test type: Superiority; p = .93, Mixed Models Analysis; Adjusted mean difference = 0.001, 95% CI 2-sided [-0.03 to 0.03]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 15 months; Test type: Superiority; p = .36, Mixed Models Analysis; Adjusted mean difference = -0.02, 95% CI 2-sided [-0.06 to 0.02]

6. Secondary Outcome: Caloric Intake
Description: Food and beverage diaries will be used to calculate daily caloric intake from foods and beverages.
Time Frame: Baseline and 7-months after the start of the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 647 | 548
kcal/day
  Total - baseline | 1636 (796) | 1699 (727)
  Total - month 7: number analyzed (Participants) | 600 | 531
  Total - month 7 | 1610 (805) | 1676 (782)
  Food - baseline | 1371 (705) | 1434 (654)
  Food - month 7: number analyzed (Participants) | 600 | 531
  Food - month 7 | 1380 (727) | 1425 (696)
  Beverage - baseline | 265 (214) | 265 (212)
  Beverage - month 7: number analyzed (Participants) | 600 | 531
  Beverage - month 7 | 229 (227) | 251 (231)
  Sugar-sweetened beverage (SSB) - baseline | 223 (205) | 223 (204)
  SSB - month 7: number analyzed (Participants) | 600 | 531
  SSB - month 7 | 190 (199) | 214 (223)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in total kcal intake from baseline to 7 months; Test type: Superiority; p = 0.70, Mixed Models Analysis — Because of skewed distributions, dietary outcomes were log-transformed and regression coefficients were exponentiated to derive the percent change in outcomes by intervention status over time; Percent difference in change = 1.4, 95% CI 2-sided [-5.3 to 8.5]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in intake of food kcal from baseline to 7 months; Test type: Superiority; p = .35, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Percent difference in change = 3.7, 95% CI 2-sided [-3.9 to 12.0]
Statistical Analysis 3: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in intake of beverage kcal from baseline to 7 months; Test type: Superiority; p = .35, Mixed Models Analysis; Percent difference in change = -10.6, 95% CI 2-sided [-29.2 to 8.8]
Statistical Analysis 4: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in SSB kcal from baseline to 7 months; Test type: Superiority; p = .18, Mixed Models Analysis; Percent difference in change = -17.5, 95% CI 2-sided [-37.8 to 9.6]

7. Secondary Outcome: Water Intake - Grams Consumed
Description: Food and beverage diaries will be used to calculate daily water intake.
Time Frame: Baseline and 7-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 647 | 548
grams/day
  Baseline | 414 (443) | 454 (441)
  Month 7: number analyzed (Participants) | 600 | 531
  Month 7 | 462 (576) | 441 (472)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change from baseline to 7 months; Test type: Superiority; p = .59, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Percent difference in change = 9.1, 95% CI 2-sided [-20.6 to 49.9]

8. Secondary Outcome: Beverage Intake
Description: Beverage intake frequency questionnaires will be used to calculate past-week frequency of beverages consumed (times per day).
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: times per day
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 677 | 572
times per day
  Water - baseline | 6.1 (4.3) | 5.7 (4.2)
  Water - month 7: number analyzed (Participants) | 639 | 556
  Water - month 7 | 7.1 (5.2) | 5.2 (3.9)
  Water - month 15: number analyzed (Participants) | 548 | 510
  Water - month 15 | 6.2 (4.7) | 4.8 (3.8)
  SSB - baseline | 3.5 (4.2) | 3.5 (4.2)
  SSB - month 7: number analyzed (Participants) | 639 | 556
  SSB - month 7 | 2.4 (3.5) | 2.8 (3.7)
  SSB - month 15: number analyzed (Participants) | 548 | 510
  SSB - month 15 | 2.1 (2.8) | 2.2 (2.9)
  Juice - baseline | 0.8 (1.1) | 0.8 (1.1)
  Juice - month 7: number analyzed (Participants) | 639 | 556
  Juice - month 7 | 0.6 (1.0) | 0.6 (0.8)
  Juice - month 15: number analyzed (Participants) | 548 | 510
  Juice - month 15 | 0.5 (1.0) | 0.5 (0.9)
  Flavored milk - baseline | 0.5 (0.9) | 0.5 (0.9)
  Flavored milk - month 7: number analyzed (Participants) | 639 | 556
  Flavored milk - month 7 | 0.4 (0.7) | 0.4 (0.8)
  Flavored milk - month 15: number analyzed (Participants) | 548 | 510
  Flavored milk - month 15 | 0.4 (0.8) | 0.4 (0.9)
  Plain milk - baseline | 1.2 (1.4) | 1.1 (1.3)
  Plain milk - month 7: number analyzed (Participants) | 639 | 556
  Plain milk - month 7 | 1.2 (1.6) | 1.0 (1.2)
  Plain milk - month 15: number analyzed (Participants) | 548 | 510
  Plain milk - month 15 | 1.1 (1.4) | 1.0 (1.2)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from baseline to 7 months; Test type: Superiority; p < .001, Mixed Models Analysis; Percent difference in change = 23.2, 95% CI 2-sided [13.1 to 34.2]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from baseline to 15 months; Test type: Superiority; p = .004, Mixed Models Analysis; Percent difference in change = 14.7, 95% CI 2-sided [4.5 to 25.9]
Statistical Analysis 3: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in SSB intake from baseline to 7 months; Test type: Superiority; p = 0.063, Mixed Models Analysis; Percent difference in change = -8.0, 95% CI 2-sided [-15.7 to 0.4]
Statistical Analysis 4: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in SSB intake from baseline to 15 months; Test type: Superiority; p = .56, Mixed Models Analysis; Percent difference in change = -2.8, 95% CI 2-sided [-11.7 to 6.9]
Statistical Analysis 5: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in juice intake from baseline to 7 months; Test type: Superiority; p = .68, Mixed Models Analysis; Percent difference in change = 1.2, 95% CI 2-sided [-4.3 to 7]
Statistical Analysis 6: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in juice intake from baseline to 15 months; Test type: Superiority; p = .66, Mixed Models Analysis; Percent difference in change = -1.4, 95% CI 2-sided [-7.4 to 5]
Statistical Analysis 7: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in flavored milk intake from baseline to 7 months; Test type: Superiority; p = 0.079, Mixed Models Analysis; Percent difference in change = -4.0, 95% CI 2-sided [-8.3 to 0.5]
Statistical Analysis 8: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in flavored milk intake from baseline to 15 months; Test type: Superiority; p = .26, Mixed Models Analysis; Percent difference in change = -3.0, 95% CI 2-sided [-8.0 to 2.3]
Statistical Analysis 9: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in plain milk intake from baseline to 7 months; Test type: Superiority; p = .20, Mixed Models Analysis; Percent difference in change = 4.4, 95% CI 2-sided [-2.2 to 11.5]
Statistical Analysis 10: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in plain milk intake from baseline to 15 months; Test type: Superiority; p = .51, Mixed Models Analysis; Percent difference in change = 2.3, 95% CI 2-sided [-4.4 to 9.6]

9. Secondary Outcome: Water Intake
Description: Direct observations of water consumed at lunchtime, 4th-grade physical education (PE) classes, and recess. Researchers tallied the number of students using water sources and the student census in the area to estimate the proportion using stations or fountains.
Time Frame: Baseline, 7-months, and 15-months after the start of the study.
Population: Data were collected from students from participating schools, whether the students were enrolled in the study, or not. For each observation type (lunchtime, PE class, and recess) and period, the number estimated in the census at each respective time point are included in the analysis. Outcome measure data were not collected from adults.
Measure: Mean (Standard Deviation); unit: observations
Arm/Group | Water Access and Promotion - Students | Control - Students
Number analyzed (Participants) | 4091 | 3947
observations
  Lunch - baseline | 3.5 (6.1) | 3.7 (6.1)
  Lunch - month 7: number analyzed (Participants) | 4019 | 3515
  Lunch - month 7 | 38.3 (15.9) | 3.6 (4.7)
  Lunch - month 15: number analyzed (Participants) | 3954 | 3936
  Lunch - month 15 | 9.2 (7.7) | 3.2 (3.1)
  Recess - baseline: number analyzed (Participants) | 1475 | 1239
  Recess - baseline | 6.5 (3.4) | 6.1 (4.5)
  Recess - month 7: number analyzed (Participants) | 1463 | 1265
  Recess - month 7 | 29.3 (36.5) | 6.6 (4.1)
  Recess - month 15: number analyzed (Participants) | 1458 | 1251
  Recess - month 15 | 8.8 (3.1) | 3.3 (3.0)
  PE class - baseline: number analyzed (Participants) | 285 | 353
  PE class - baseline | 66.6 (87.8) | 47.4 (32.2)
  PE class - month 7: number analyzed (Participants) | 272 | 284
  PE class - month 7 | 89.6 (58.7) | 53.2 (65.6)
  PE class - month 15: number analyzed (Participants) | 271 | 307
  PE class - month 15 | 95.0 (56.2) | 43.1 (38.1)
Statistical Analysis 1: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from water source at lunch from baseline to 7 months; Test type: Superiority; p < .001, Mixed Models Analysis; Percent difference in change = 31.3, 95% CI 2-sided [21.2 to 42.2]
Statistical Analysis 2: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from water source during lunch from baseline to 15 months; Test type: Superiority; p = .22, Mixed Models Analysis; Percent difference in change = 4.9, 95% CI 2-sided [-3.0 to 13.5]
Statistical Analysis 3: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from water source at recess from baseline to 7 months; Test type: Superiority; p = .02, Mixed Models Analysis; Percent difference in change = 17.0, 95% CI 2-sided [2.6 to 33.3]
Statistical Analysis 4: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from water source at recess from baseline to 15 months; Test type: Superiority; p = .48, Mixed Models Analysis; Percent difference in change = 4.7, 95% CI 2-sided [-8.0 to 19.2]
Statistical Analysis 5: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from water source at PE from baseline to 7 months; Test type: Superiority; p = .14, Mixed Models Analysis; Percent difference in change = 34.6, 95% CI 2-sided [-9.4 to 99.8]
Statistical Analysis 6: Comparison: Water Access and Promotion - Students vs Control - Students; Analysis of between group change in water intake from water source at PE from baseline to 15 months; Test type: Superiority; p = .16, Mixed Models Analysis; Percent difference in change = 32.1, 95% CI 2-sided [-11.0 to 96.2]

10. Other Pre Specified Outcome: School Policies and Practices
Description: School administrators and food service director surveys of nutrition and physical activity policies and practices at schools
Time Frame: Baseline and 15-months after the start of the study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Water Access and Promotion - Students | Water Access and Promotion - School Personnel | Control - Students | Control - School Personnel | Food Service Directors
All-Cause Mortality (participants affected / at risk) | 1/680 | 0/10 | 0/582 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/680 | 0/10 | 0/582 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/680 | 0/10 | 0/582 | 0/12 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Water Access and Promotion - Students (N=680) | Water Access and Promotion - School Personnel (N=10) | Control - Students (N=582) | Control - School Personnel (N=12) | Food Service Directors (N=13)
Death (General disorders) | 1 | 0 | 0 | 0 | 0 — Cause of death not disclosed to research team due to privacy concern

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03181971/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03181971/SAP_001.pdf
  • Informed Consent Form (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03181971/ICF_002.pdf